CLINICAL TRIAL: NCT02700802
Title: Mitigating Hunger and Food Insecurity Among Socioeconomically Disadvantaged Caregivers of Hospitalized Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This research described in this protocol was not funded.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB16-1434
Record Dates: First submitted 2016-03-01; First posted 2016-03-07 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Health Behavior
Keywords: food insecurity; informal caregiver health; clinic-to-community linkages; community resources
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Feed1st: Face-to-face provider delivered referral (Experimental): In this arm of the study, caregivers will receive usual care and a brief face-to-face referral to the Feed1st program delivered by the provider.
  Interventions: Other: Feed1st
- Feed1st: Text message delivered referral (Experimental): In this arm of the study, caregivers will receive usual care and an automated brief text message referral to the Feed1st program from the health care provider. The text message referral will align as closely as possible with the face-to-face referral.
  Interventions: Other: Feed1st
- Standard of Care (No Intervention): Usual care includes passive delivery of information from nursing staff about all available food options in the hospital including the self-serve food pantries in the standard Caregiver FYI Admissions Packet.

INTERVENTIONS:
Other: Feed1st — Feed1st is a unique hospital-based hunger mitigation program that, since 2010, has operated low-cost, self-serve food pantries at Comer Children's Hospital. All parents and caregivers with a hospitalized child have 24/7 free access to these self-serve pantries with the option to eat food in the pantry, carry out as much food as needed, and contribute back to the pantry with food, volunteerism, or other resources. The program also offers free phone/text/email navigation for food support and other basic needs resources. We aim to conduct a 3-arm, randomized comparative effectiveness study to evaluate the impact, versus usual care, of two alternative referral strategies to increase Feed1st program utilization and impact.
  Arms: Feed1st: Face-to-face provider delivered referral; Feed1st: Text message delivered referral

SUMMARY:
The Feed1st proposed program of research will promote health of informal caregivers with a hospitalized child by testing a self-management intervention that addresses the widely overlooked problem of caregiver hunger. As many as 54% of parents and other informal caregivers of hospitalized children struggle with insufficient food to nourish themselves and their family during and after a hospital stay. Hunger impairs caregiver physical and mental health by depleting energy for self-care, emotional self-regulation, and supportive interactions with the child, the family, and the formal caregiver team. The long-term objective of the Feed1st program is to alleviate hunger and food insecurity among families with hospitalized children. Established in partnership with nursing and chaplaincy leadership at our children's hospital and the Greater Chicago Food Depository, the Feed1st program currently operates self-serve food pantries on four inpatient units and the emergency department in our children's hospital on Chicago's South Side. Since 2010, Feed1st has provided nearly 8500 pounds of food to at least 4,000 individuals and 1500 households via the self-serve food pantries in the children's hospital. Over this same period, our team has also created a system for efficiently connecting families to community-based resources for hunger and other basic needs.

ELIGIBILITY:
Inclusion Criteria:

- 18 years of age or older and English speaking, the primary caregiver to a dependent child younger than age 18, have been screened for household food insecurity, reside in the 16 zip code primary service area geography,

Exclusion Criteria:

* Caregivers of children in the neonatal intensive care unit (NICU) will be excluded to minimize infectious risk to critically ill newborns and their caregivers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in mental health-related quality of life at 6 months | Baseline, 4-7 days, 3 months, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stacy T Lindau, MD, MAPP, Principal Investigator — University of Chicago